CLINICAL TRIAL: NCT05179655
Title: TEENS Multi-site Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Region of Southern Denmark (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Britt Reuter Morthorst, Associate Professor, Senior researcher, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-21035306
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-11

CONDITIONS: Self-Injurious Behavior
Keywords: Internet-based intervention; Online therapy; Emotion regulation; ERITA
MeSH Terms: conditions — Self-Injurious Behavior; Emotional Regulation | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: An investigator-initiated, multi-site randomised, parallel group, clinical superiority trial with blinded outcome assessment investigating the internet-based intervention ERITA as add-on to TAU compared to TAU alone in NSSI engaging psychiatric, outpatient youth. Participants will be randomised at the allocation ratio 1:1. Randomisation will be handled centrally at the Copenhagen Trial Unit (CTU) using a computer-generated allocation sequence with a varying block size concealed from the investigators. The allocation sequence will be stratified NSSI at baseline 1-10 versus 11≤ episodes in the past month, and trial site. CTU will generate the allocation sequence and investigators at the clinical trial sites will assign participants to the intervention groups using an OpenClinica web-based system developed by the CTU
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, a blinding of participants and therapists is not possible. Blinded outcome assessment will be performed by a trained researcher. Statistical analyses will be performed by two blinded statisticians presenting independent reports and with the intervention groups coded as A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERITA + TAU (Treatment as usual) (Experimental): The Emotion Regulation Individual Therapy for Adolescents (ERITA) intervention as add-on to TAU consists of 11 weeks, manualized online therapy based on the methods of Cognitive Behavioral Therapy (CBT), Dialectical Behavior Therapy (DBT), and Acceptance and Commitment Therapy (ACT) adapted for youth
  Interventions: Behavioral: Emotion Regulation Individual Therapy for Adolescents (ERITA); Other: Treatment as usual
- TAU (Treatment as usual) (Other): Within mental health services in Denmark child and adolescent psychiatrists provide specialized treatment for young psychiatric patients as outpatient services. In this study the control intervention (TAU) consists of clinical assessment and treatment for patient's current primary psychiatric condition (referral condition and A-diagnosis).
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Emotion Regulation Individual Therapy for Adolescents (ERITA) — The ERITA intervention as add-on to TAU consists of 11 weeks, manualized online therapy based on the methods of Cognitive Behavioral Therapy (CBT), Dialectical Behavior Therapy (DBT), and Acceptance and Commitment Therapy (ACT) adapted for youth. The ERITA content consists of psychoeducation, emotion recognition, awareness training and theory of emotion regulation, including acceptance and validation skills.
  Other Names: ERITA
  Arms: ERITA + TAU (Treatment as usual)
Other: Treatment as usual — Within Mental Health Services in Denmark child and adolescent psychiatrists provide specialized treatment for young psychiatric patients as outpatient services. In this trial the control intervention is treatment as usual (TAU) and consists of clinical assessment and treatment for patient's current primary psychiatric condition. TAU encounters a variety of clinical treatment and assessment offers, however, all within the field of expertise in child and adolescent psychiatry; out-patient care may consist of treatment for OCD, eating disorders, psychoses or affective disorders. TAU may consist of pharmacological treatment, Family-Based Treatment (FBT), Cognitive Behavioral Therapy (CBT), supportive counselling and/or psychoeducation.

SUMMARY:
Emotion Regulation Individual Therapy for Adolescents, also called ERITA, is a youth friendly online therapy aiming to provide skills and train emotion regulation.

The aim of the TEENS Multi-site Trial is to investigate the effect of ERITA, including an app, as add-on to treatment as usual in young patients referred to Mental Health Services. We expect 356 families to participate from three designated Regions in Denmark.

DETAILED DESCRIPTION:
Background: A prevalence of non-suicidal self-injury is not easily assessed; however, meta-analyses found a lifetime prevalence of 17% in non-clinical student samples. This estimate increases to 50-74% in psychiatric populations. Non-suicidal self-injury is an important predictor for later suicidal behavior and death by suicide. Although non-suicidal self-injury is highly prevalent, there is no evidence for specific treatment for non-suicidal self-injury in adolescents. Reviews find that internet-based interventions guided by a therapist are effective for several psychiatric disorders such as anxiety and depression in adult population. Patients with stigmatizing illnesses such as non-suicidal self-injury may be reluctant to seek help and adhere with treatment while internet-based interventions are more appealing. There is a need for trials investigating the effect of specialized interventions for non-suicidal self-injury in youth, including digital interventions.

Objective: To investigate the effect of an internet-based intervention, Emotion Regulation Individual Therapy for Adolescents (ERITA), as add-on to treatment as usual in 13-17-year-old patients with non-suicidal self-injury referred to Child- and Adolescent Mental Health Services with subsequent non-suicidal self-injury as primary outcome assessed by Deliberate Self-Harm Inventory - Youth. Further clinical outcomes such as quality of life, depression, anxiety and stress, as well as emotion regulation difficulties will be assessed as secondary outcomes.

Method and materials: This is a randomized, clinical, superiority, multicenter trial in a parallel group design. Patients will be recruited from Child- and Adolescent Mental Health Services in three of the Danish Regions: The trial inclusion period will be from primo 2022 to ultimo 2023. The experimental intervention is therapist guided internet-based ERITA provided exclusively online as add-on to treatment as usual in the experimental group. Treatment as usual is provided by multidisciplinary teams in outpatient clinics in all participating regions. We expect to include 356 participants and one of their parents.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 5 non-suicidal self-injury episodes in the past year and ≥ 1 non-suicidal self-injury episodes in the past month assessed by the Deliberate Self-Harm Inventory, Youth version (DSHI-Y).
* Age-appropriate literacy assessed by referring clinicians and the self-injury team, i.e. age between 13 and 17.
* Having at least one parent committing to participate in the parent program.
* Informed consent from parents/legal caretakers and assent from participants above 15 years of age.

Exclusion Criteria:

* Imminent suicidal risk assessed by clinicians during routine screening procedure (that can be rated as no risk, elevated risk, or imminent risk) in need of admission or other life saving strategies.
* Lack of informed consent from parents/legal caretakers.
* Lack of informed assent from the participant above 15 years of age.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 356 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-suicidal self-injury episodes | End of treatment after 12 weeks and 6 months follow-up
  Non-suicidal self-injury within the last four weeks, at end of intervention (12 weeks) by blinded outcome assessment by phone or video conference measured by Deliberate Self-Harm Inventory

SECONDARY OUTCOMES:
Kidscreen-10; Quality of life | End of treatment after 12 weeks and 6 months follow-up
  Quality of life at 12 weeks, assessed with Kidscreen-10, a five point likert scale, range: not at all, a little, moderate, much, very much.
Symptoms of depression, anxiety and stress | End of treatment after 12 weeks and 6 months follow-up
  Symptoms of depression, anxiety and stress at 12 weeks, assessed with Depression Anxiety Stress Scale (DASS-21) presented as analyses for each subgroup item. Four point likert scale, range: did not apply to me, applied to me to some degree, applied to me to a considerable degree, applied to me much/most of the time. Total rage for subscores: 0-42. Higher scores reflect worse outcome.
Non-suicidal self-injury as dichotomous (any/none) | End of treatment after 12 weeks and 6 months follow-up
  The proportion of participants with any NSSI during the past four weeks.

OTHER OUTCOMES:
Difficulties in emotion regulation | End of treatment after 12 weeks and 6 months follow-up
  Difficulties in emotion regulation, assessed with Difficulties in Emotion Regulation Scale - 16 Item Version (DERS-16). DERS-16 has 16 items which each generates a score from 1 to 5. The results will be presented as one sum-score. The scores in this scale range from 16-80 with higher scores indicating greater emotion regulation difficulties.
Borderline Symptom List (BSL-supplement). | Through trial periode (every three weeks, end of treatment after 12 weeks and 6 months follow-up)
  Indirect self-destructive behaviours assessed with Borderline Symptom List (BSL-supplement). BSL-supplement has 11 items which each generates a score from 0 to 4. The results will be presented as one sum-score.
Suicidal ideations | Through trial period (every three weeks, end of treatment after 12 weeks and 6 months follow-up)
  Suicidal ideations assessed by SIDAS. A five item scale with questions ranging from 0 to 10. Final sum score from 0-50.
Coping with Children's Negative Emotions - Adolescents | End of treatment after 12 weeks and 6 months follow-up
  Adolescent rated parents' ability to cope with children's negative emotions assessed with The Coping with Children's Negative Emotions Scale (CCNES-APP). 9 main items with 6 sub items (a to f) for each. Each sub item generates a score from 1 to 7. The results will be presented as mean-scores for the six subscales.
Coping with Children's Negative Emotions - Parents | End of treatment after 12 weeks and 6 months follow-up
  Parent-rated perceived ability to cope with children's negative emotions assessed with The Coping with Children's Negative Emotions Scale Adolescent (CCNES-A). 9 main items with 6 sub items (a to f) for each. Each sub item generates a score from 1 to 7. The results will be presented as mean-scores for the six subscales.
Negative Effects Questionnaire | Through trial periode (every three weeks and end of treatment after 12 weeks)
  Adverse Events of therapy assessed with Negative Effects Questionnaire (NEQ). NEQ has 20 items, with 5 sub-items The results will be presented as means and standard deviations.
Working Alliance | Through the trial period (week four and eight)
  The alliance percieved between the participant and the therapist, WAI-SR

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Pagsberg, Professor, Study Chair — Mental Health Services Capital Region Denmark
Locations (4):
- Denmark (4):
  - Child and Adolescent Mental Health Services, Aalborg
  - Child and Adolescent Mental Health Services Southern Region Denmark, Odense
  - Child and Adolescent Mental Health Services in Region Zealand, Roskilde
  - Team for Self-injury, Child and Adolescent Mental Health Services, B195, Copenhagen, Ø